CLINICAL TRIAL: NCT03608982
Title: Evaluating the Impact of Simulated Patients on Knowledge, Skills and Attitudes of Laypeople Following a Basic First-Aid Course: A Cluster-Randomized Controlled Trial
Brief Title: The Use of Simulated Patients During Basic-first Aid Courses for Laypeople
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Evidence-Based Practice, Belgium (Other)
Collaborators: Belgian Red Cross (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SIM-001; G- 2018 06 1273 (Other: Social Medical Ethical Comission (SMEC) of KU Leuven)
Record Dates: First submitted 2018-07-05; First posted 2018-08-01 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Burns; Stroke
Keywords: First aid; Simulated patient; Laypeople
MeSH Terms: conditions — Burns; Stroke

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized trial, in which allocation is done at the level of the companies that request a first aid course for their employees.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed about participating in a study, evaluating the performance of basic first aid courses taught by the Belgian Red Cross, but will be blinded from the actual goal of the research, i.e. testing the added value of simulated patients.
  The outcome assessors will not be aware of the allocation status of participants whose practical skills they judge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulated patient (Experimental): The materials in this course are standardized, and consist of lectures with a slide show, questions & answers conversations, and practical exercises on fellow-students. The courses are being taught by professional first aid tutors from the Belgian Red Cross. During the practical exercises, a simulated patient will unexpectedly enter the room requiring treatment.
  Interventions: Other: Simulated patient
- No simulated patient (Active Comparator): The course materials in the control courses are also standardized. Instead of using simulated patients, however, video clips will be shown to demonstrate the first aid techniques.
  Interventions: Other: No simulated patient

INTERVENTIONS:
Other: Simulated patient — The simulated patient is a professional actor and Belgian Red Cross employee, who combines acting distress and pain with moulage, to mimic the injuries as truthfully as possible. For feasibility reasons, the simulant will only be included in two sections of the course: the respective treatments of burns and stroke. The remainder of the course will be taught without simulated patient by the professional first aid tutors.
  Arms: Simulated patient
Other: No simulated patient — Instead of a simulated patients, participants get to watch video clips on first aid techniques.
  Arms: No simulated patient

SUMMARY:
Background: Teaching first aid to laypeople is a cost-effective way to improve public health. However, it is currently unclear what the most effective ways are to teach first aid. It has already been shown that simulated patients have an added value in teaching emergency care to healthcare professionals.

This paper describes the protocol for a cluster-randomized controlled trial that will investigate the influence of using a simulated patient during basic first aid training for laypeople on laypeople's knowledge, skills and self-efficacy.

Hypothesis: The null hypothesis of this research is that the use of simulated patients during basic first aid training does not result in a statistically significant change in knowledge, skills and self-efficacy concerning the first aid topics for which a simulated patient is used. The alternative is that knowledge, skills and self-efficacy will be influenced by using simulated patients.

Methods: This study will be a cluster-randomized controlled trial, that will take place from September 2018 to June 2020. The study population will consist of employees taking a three day first aid certification course with the Belgian Red Cross. The employers requesting a first aid course will be randomised in receiving a course with or without simulated patient. The simulated patient will only be used for the topics first aid for burns and first aid for stroke in the intervention group. The participants will complete a questionnaire to measure their knowledge and self-efficacy before and after the course, and complete a practical skills test after the course testing these first aid topics. To test whether the retention of first aid knowledge and self-efficacy is influenced by using a simulated patient during a certification course, participants following a refresher course one year after the certification course will complete a follow-up questionnaire.

This cluster-randomized controlled trial will be, to the investigator's knowledge, the first to investigate the added value of simulated patients during first aid courses for laypeople.

ELIGIBILITY:
Inclusion Criteria:

* Employed in a company requesting a basic first aid course taught by the Belgian Red Cross

Exclusion Criteria:

* Employed in a company that purposefully requests a simulated patient
* Employed in a company that requests a course in a language other than Dutch (French, English)
* Participants < 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1168 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in first aid knowledge, measured as the change in average score on a questionnaire of 10 questions (multiple choice) related to first aid topics for which a simulated patient was used during the basic first aid course. | At the start of the basic first aid course and at one year follow-up, right before the participants follow their yearly refresher course (between 10 months and 14 months after the basic first aid course).
  10 multiple choice questions testing knowledge concerning first aid for burns and stroke, blended in with 10 questions for other first aid topics for the purpose of blinding the participants
First aid skills, measured during a practical skills test evaluating a total of 14 skills concerning the first aid topics for which a simulated patient was used during the basic first aid course | At the end of the basic first aid course, during the evaluation moment in the afternoon of the final day of the three-day course.
  Practical skills concerning first aid for burns and stroke, blended in with practical skills tests for cardiopulmonary resuscitation and two other first aid topics for the purpose of blinding the participants.
Change in first aid self-efficacy, measured as the change in average score on a questionnaire of 6 questions (5-point Likert scale), related to first aid topics for which a simulated patient was used during the basic first aid course. | At the start of the basic first aid course and at one year follow-up, right before the participants follow their yearly refresher course (between 10 months and 14 months after the basic first aid course).
  6 questions to be answered on a 5-point Likert scale, testing self-efficacy concerning first aid for burns and stroke, blended in with 6 questions concerning self-efficacy for other first aid topics for the purpose of blinding the participants.

SECONDARY OUTCOMES:
Change in first aid knowledge, measured as the change in average score on a questionnaire of 10 questions (multiple choice) related to first aid topics for which a simulated patient was used during the basic first aid course. | At the start of the basic first aid course and at the end of the basic first aid course, during the evaluation moment in the afternoon of the final day of the three-day course.
  10 questions testing knowledge concerning first aid for burns and stroke, blended in with 10 questions for other first aid topics for the purpose of blinding the participants.
Change in first aid self-efficacy, measured as the change in average score on a questionnaire of 6 questions (5-point Likert scale), related to first aid topics for which a simulated patient was used during the basic first aid course. | At the start of the basic first aid course and at the end of the basic first aid course, during the evaluation moment in the afternoon of the final day of the three-day course..
  6 questions to be answered on a 5-point Likert scale, testing self-efficacy concerning first aid for burns and stroke, blended in with 6 questions concerning self-efficacy for other first aid topics for the purpose of blinding the participants.
Participant's satisfaction with the basic first aid course provided, measured using a 10-point scale | At the end of the basic first aid course, during the evaluation moment in the afternoon of the final day of the three-day course.
  Participant's general satisfaction concerning the basic first aid course they received will be verified using a 10-point scale (ranging from 1: not satisfied at all to 10: very satisfied).
Costs | At the start of the basic first aid course, immediately after the basic first aid course, during the evaluation moment, and at one year follow-up, right before the participants follow their yearly refresher course (between 10 months and 14 months)
  Costs associated with a course, relatively to the gain in knowledge and self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Emmy De Buck, Phd, Principal Investigator — Centre for Evidence-Based Practice, Belgium
Locations (1):
- Belgian Red Cross, Mechelen, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Avau B, Vanhove AC, Vandenlindenloof M, Suls L, Verstraeten H, Vandekerckhove P, De Buck E. Evaluating the Impact of Simulated Patients on Knowledge, Skills and Attitudes of Laypeople Following a Basic First Aid Course: Protocol for a Cluster-Randomized Controlled Trial. International Journal of First Aid Education 2019, Vol. 2 Issue 2, Article 3.
- [Result] Avau B, Vanhove AC, Scheers H, Stroobants S, Lauwers K, Vandekerckhove P, De Buck E. Impact of the Use of Simulated Patients in Basic First Aid Training on Laypeople Knowledge, Skills, and Self-efficacy: A Controlled Experimental Study. Simul Healthc. 2022 Aug 1;17(4):213-219. doi: 10.1097/SIH.0000000000000657. Epub 2022 Apr 5. PMID 35921627